CLINICAL TRIAL: NCT06054178
Title: Intraoperative Nerve Identification With Fluorescein Sodium
Brief Title: Identification of Nerves Using Fluorescein Sodium
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Tulio Valdez, Professor of Otolaryngology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 71857; R25DC020174-03 (NIH)
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Pleomorphic Adenoma of the Parotid; Warthin Tumor; Head and Neck Disorder; Head and Neck; Thyroid Disease; Thyroidectomy
MeSH Terms: conditions — Adenolymphoma; Thyroid Diseases | interventions — Fluorescein

STUDY DESIGN:
Intervention Model Description: Experimental: Fluorescein sodium during surgery
  Subjects undergoing parotid surgery for benign conditions will have fluorescein sodium administered intravenously after induction, and fluorescence imaging will be performed to visualize nerves intraoperatively
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fluorescein sodium during surgery (Experimental): Subjects undergoing parotid surgery for benign conditions will have fluorescein sodium administered intravenously after induction, and fluorescence imaging will be performed to visualize nerves intraoperatively
  Interventions: Drug: Fluorescein Sodium

INTERVENTIONS:
Drug: Fluorescein Sodium — Intravenous administration of 1 mg/kg. If initial dosing is insufficient, additional doses may be administered up to a total of 3 mg/kg
  Other Names: FLUORESCITE Injection 10%

SUMMARY:
The purpose of this study is to see if there is benefit in using an IV contrast (sodium fluorescein) to identify nerves during head and neck surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects
2. 18 years or older
3. Scheduled for open head and neck surgery

Exclusion Criteria:

1. Inability or unwillingness of a subject
2. Pregnancy
3. Vulnerable or disadvantaged population (pregnant women, decisionally impaired, homeless, employees, students)
4. Patients with severe medical condition(s) that in the view of the investigator prohibits participation in the study
5. History of adverse reaction to fluorescein including allergy.
6. History of renal failure or chronic kidney disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Facial nerve correlation of Fluorescein Sodium With Electrostimulation | Intraoperative
  Surgeon assessment of fluorescence correlation with electrostimulation using a Likert-style rating from 1-4 where 1=No correlation; 2=Some correlation; 3=Good correlation; 4=Excellent correlation
Correlation of Fluorescein Sodium With Surgeons' Visual Assessment of nerve | Intraoperative
  Survey of surgeon visual assessment of nerve under white light compared to fluorescence using a Likert-style rating from 1-4 where 1=No correlation; 2=Some correlation; 3=Good correlation; 4=Excellent correlation.
Ratio of Nerve Fluorescence compared to Background Tissue | Intraoperative
  Ratio of nerve fluorescence intensity compared to background fluorescence intensity

SECONDARY OUTCOMES:
Average Dose of Sodium Fluorescein Administration | Intraoperative
  Average dose of sodium fluorescein administered in mg/kg
Time to Nerve Visualization | Intraoperative
  Amount of time (in minutes) to nerve fluorescence after sodium fluorescein adminstration

CONTACTS AND LOCATIONS:
Overall Officials: Tulio Valdez, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Medical Center, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park RK, Arus BA, Lee JY, Weitzenberg MM, Lee MC, Nyaeme MS, Barthel J, Balsamo G, Baik FM, Speirs K, Blume B, Heller-Algazi M, Chmyrov A, Plettenburg O, Megwalu UC, Weitz J, Distler M, Bruns OT, Valdez TA. Intraoperative nerve imaging with sodium fluorescein. medRxiv [Preprint]. 2025 Feb 17:2025.02.08.25321923. doi: 10.1101/2025.02.08.25321923. PMID 40034788